CLINICAL TRIAL: NCT03428984
Title: A Phase 1, Open-Label Study to Evaluate the Safety and Pharmacokinetics of EXPAREL When Administered for Postsurgical Analgesia in Subjects Undergoing Posterolateral Thoracotomy
Brief Title: Study in Adult Subjects Undergoing Posterolateral Thoracotomy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow study enrollment
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-118
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EXPAREL 20 + 20 (Experimental): 20 mL EXPAREL with 20 mL normal saline
  Interventions: Drug: EXPAREL
- EXPAREL 20 + 10 (Experimental): 20 mL EXPAREL with 10 mL normal saline
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL — EXAPREL 266 mg in 20 mL

SUMMARY:
Primary Objective: To characterize the pharmacokinetic (PK) profile of EXPAREL when administered as a posterior intercostal nerve block.

Secondary Objective: To assess the safety and tolerability of EXPAREL in this surgical model.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label study designed to evaluate the safety and PK profile of EXPAREL when administered as a posterior intercostal nerve block. Twenty-four adult subjects undergoing thoracotomy are planned for enrollment.

Subjects will be screened within 30 days prior to study drug administration. During the screening visit, which must take place at least 1 day prior to surgery, subjects will be assessed for past or present neurologic, cardiac, and general medical conditions that, in the opinion of the investigator, would preclude them from study participation.

Subjects will undergo their pre-planned thoracotomy procedure per the institution's standard of care. Prior to wound closure, subjects will be given either 40 mL of study drug (20 mL EXPAREL expanded with 20 mL normal saline) or 30 mL of study drug (20 mL EXPAREL expanded with 10 mL normal saline). Subjects will remain in the hospital for a minimum of 48 hours for pharmacokinetic testing and evaluation of safety.

On Day 14, the subject will complete the study via phone call in order to collect safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age.
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
3. Scheduled to undergo chest surgery using either minimally invasive (VATS or robotic-assisted surgery) or open techniques (posterolateral, lateral, or anterior thoracotomy or requiring insertion of an inter-rib spreader/retractor) for a primary thoracic non-infectious indication under general anesthesia.
4. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration. Female subjects must be surgically sterile, at least 2 years menopausal, or using an acceptable method of birth control. If of childbearing potential, the subject must have a documented negative pregnancy test within 24 hours before surgery.
2. Prior ipsilateral thoracotomy (the likely presence of adhesions will limit ability to perform a precise block guided by thoracoscopy). Note: previous VATS or robotic surgery is permissible.
3. Any planned pleurodesis as part of the surgical procedure.
4. Redo ipsilateral thoracotomy
5. Received bupivacaine or any other local anesthetic within 7 days of screening.
6. Body weight < 50 kilograms (110 pounds) or a body mass index ≥ 35 kg/m2.
7. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics or opioids.
8. Previous participation in a liposome bupivacaine study.
9. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
10. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance.
11. Significant medical conditions (including widely disseminated metastatic disease) or laboratory results that, in the opinion of the investigator, indicate an increased vulnerability to study drugs and procedures.
12. History of coronary or vascular stent placed within the past 3 months (may be extended to 1 year if medically indicated per physician discretion).
13. Have been treated for a deep vein thrombosis, pulmonary embolism, myocardial infarction, or ischemic stroke within the past 6 months (may be extended to 1 year if medically indicated per physician discretion).
14. Severely impaired renal or hepatic function (eg, serum creatinine level > 2 mg/dL [176.8 μmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN], or serum alanine aminotransferase [ALT] level > 3 times ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
AUC of EXPAREL concentration | 0-72 hours
  Area under the concentration curve for EXPAREL

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | 0-14 days
  Incidence to treatment-emergent adverse events through 14 days

CONTACTS AND LOCATIONS:
Overall Officials: David Rice, MD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States